CLINICAL TRIAL: NCT04535154
Title: Patient-reported Outcomes and Lung Function After Hospitalization for COVID-19
Acronym: PROLUN
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Akershus (Other)
Collaborators: Oslo University Hospital (Other); Ostfold Hospital Trust (Other); Haukeland University Hospital (Other); St. Olavs Hospital (Other); The National Association for Heart and Lung Disease, Jessheim, Norway (Other)
Responsible Party: Principal Investigator, Gunnar Einvik, Primary Investigator, University Hospital, Akershus
Other Study IDs: PROLUN
Record Dates: First submitted 2020-08-29; First posted 2020-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Covid19; Lung Function Decreased
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No interventions — No interventions

SUMMARY:
A multicenter prospective cohort study performed at 6 major teaching hospitals in Southern Norway to study patient reported outcomes, lung function and pulmonary CT in patients at 3 and 12 months after hospitalization for coronavirus disease 2019 (COVID-19).

DETAILED DESCRIPTION:
This cohort study aim to describe the Natural course of COVID-19 disease in an consecutive and unselected cohort of Norwegians that have been hospitalized.

In addition to the primary and secondary outcomes related to PROMS, lung function and pulmonary CT, the study also have several substudies: Cardiology: The study includes echocardiography, 24-h electrocardiography and cardiopulmonary exercise test.

ENT: The study includes CT of head sinuses and patient-reported sleep disturbances and nose symptoms in a subgroup of patients.

Laboratory: Analyses of common markers of inflammation and cardiac biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Discharged before June 1 2020 after hospitalization at participating hospital for COVID-19

Exclusion Criteria:

* Age < 18 years
* Dementia
* Living outside hospital catchment area
* Participation in WHO COVID-19 clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients hospitalized who have been hospitalized for COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 264 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Forced vital capacity | 3 months
  L
Forced vital capacity | 12 months
  L
Gas diffusion capacity of carbon monoxide | 3 months
  mmol/kPa*min
Gas diffusion capacity of carbon monoxide | 12 months
  mmol/kPa*min
modified Medical Respiratory Council Dyspnea Scale | 6 weeks
  Unit
modified Medical Respiratory Council Dyspnea Scale | 3 months
  Unit
modified Medical Respiratory Council Dyspnea Scale | 12 months
  Unit
Parenchymal opacities of the lungs | 3 months
  Number of opacities in one lung zone
Parenchymal opacities of the lungs | 12 months
  Number of opacities in one lung zone

SECONDARY OUTCOMES:
Forced expiratory capacity during 1st second of expiration | 3 months
  L
Forced expiratory capacity during 1st second of expiration | 12 months
  L
FEV1/FVC | 3 months
  Percentage
FEV1/FVC | 12 months
  Percentage
Gas diffusion capacity adjusted for alveolar ventilation (KCO) | 3 months
  mmol/kPa*min*L
Gas diffusion capacity adjusted for alveolar ventilation (KCO) | 12 months
  mmol/kPa*min*L

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Einvik, PhD, Principal Investigator — University Hospital, Akershus
Locations (1):
- Dept Pulmonary Medicine, Lørenskog, Akershus, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ingul CB, Grimsmo J, Mecinaj A, Trebinjac D, Berger Nossen M, Andrup S, Grenne B, Dalen H, Einvik G, Stavem K, Follestad T, Josefsen T, Omland T, Jensen T. Cardiac Dysfunction and Arrhythmias 3 Months After Hospitalization for COVID-19. J Am Heart Assoc. 2022 Feb;11(3):e023473. doi: 10.1161/JAHA.121.023473. Epub 2022 Jan 20. PMID 35048715

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-22): https://cdn.clinicaltrials.gov/large-docs/54/NCT04535154/Prot_SAP_000.pdf